CLINICAL TRIAL: NCT06446687
Title: Radiographic Assessment of Bone Gain Following Sinus Lifting With Simultaneous Implant Placement Using Crestal Approach With Membrane Control Technique for Bone Augmentation of Atrophied Maxillary Posterior Ridge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Hadi Homoud Radi, Affiliation oral and maxillofacial surgery master candidate at cairo university, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99522504
Record Dates: First submitted 2024-05-13; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Implant Site Reaction; Maxillary Deficiency
Keywords: Closed Sinus lifting; Bone Gain
MeSH Terms: conditions — Retrognathia | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sinus Lifting by Using Crestal approach with membrane control technique. (Experimental): Sinus Lifting with simultaneously implant placement.
  Interventions: Procedure: Dental implant with sinus lifting.

INTERVENTIONS:
Procedure: Dental implant with sinus lifting. — Surgery will be performed under local infiltration anaesthesia. Flap will be done. For maxillary sinus lifting by using Crestal approach with Membrane Control Technique by Wang (Wang, 2017) will be employed. After reflecting on the flap, Magic Split will be used to confirm bone quality clinically. This will be followed by site preparation using Magic Marking Drill. Bone drilling will then be performed by Magic Drill shorter by 2 mm from the sinus floor. This will be followed by sinus lifting by using Magic Sinus Lifter (MSL). The 3mm space of the apex of the Sinus Lifter instrument enables direct control of the bone-block and consequently the membrane, which is connected to the bone-block. the fixture will be installed in the conventional method. Then cover the fixture with the cover screw. The flap will be sutured. An immediate CBCT will be requested to ensure the implant is in its proper position.

SUMMARY:
This study aims to evaluate the quantity and quality of the native and the newly bone around dental implants that's simultaneously installed with sinus lifting

ELIGIBILITY:
Inclusion Criteria:

1. Patients required dental implant treatment in the posterior maxilla, in the premolar and molar regions ( both sexes).
2. Residual bone height 4-8mm in the estimated implant positions.
3. The bone width of the alveolar ridge is at least 5mm in estimated implant positions.
4. The edentulous ridges are covered with optimal thickness of mucoperiosteum.

Exclusion Criteria:

1. Patients with a systemically diseases or inflammation whether local or generalized.
2. Patients with bleeding disorders.
3. Subjected to irradiation in the head and neck area less than 1 year before implantation.
4. Poor oral hygiene and motivation.
5. Pregnant or nursing.
6. Severe bruxism or clenching.
7. Active infection or severe inflammation in the area intended for implant placement.
8. Unable to open mouth sufficiently to accommodate the surgical tooling.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Cone beam computed tomography (CBCT) bone height formation around dental implants | Patients will be evaluated after 3 days and weekly for the first month and then once monthly up to 4 months for signs of dehiscence. then cone-beam computed tomography 4 months postoperatively to calculate the amount of vertical bone gain.
  Calculate bone height and formation around dental implants.

SECONDARY OUTCOMES:
Cone beam computed tomography (CBCT) density formation around dental implants | Patients will be evaluated after 3 days and weekly for the first month and then once monthly up to 4 months for signs of dehiscence. then cone-beam computed tomography 4 months postoperatively to calculate the amount of vertical bone gain.
  Calculate bone density formation around dental implants.

IPD SHARING:
Plan to Share IPD: No